CLINICAL TRIAL: NCT03387865
Title: A Clinico-biological Database of Lung Cancers
Acronym: Bio-lung
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Lille (Other)
Collaborators: Institut Pasteur de Lille (Other); University of Lille Nord de France (Other)
Responsible Party: Sponsor
Other Study IDs: 2015_43; 2016-A01383-48 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2017-11-21; First posted 2018-01-02 (Actual); Last update posted 2022-10-19 (Actual); Status verified 2022-10

CONDITIONS: Lung Cancer
Keywords: banking, biological sampling, tumor tissue, tumor response
MeSH Terms: conditions — Lung Neoplasms; Neoplasms | interventions — Blood Specimen Collection; Gene Library

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — serum, plasma, tumor tissue, healthy tissue, stools (gut microbiome)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: tissue biopsies — additional biopsies will be performed during a diagnostic or therapeutic procedure, in order to sample tumor tissue and healthy tissue.
Procedure: blood sampling — additional blood samples will be collected during a SOC sampling procedure (2 EDTA 7.5 ml tubes, 2 SST 7.5 ml tubes and 2 citrate 5 ml tubes)
Genetic: DNA banking — constitutional and somatic genetic alterations will be analysed for subjects who consent, from either tumor or healthy tissue, or whole blood buffy coat after centrifugation

SUMMARY:
This prospective, single-center, interventional study is conducted in order to achieve a biological bank accompanied by clinical data. Blood samples, optional tumor tissue and fecal samples are collected, processed and banked for all the included subjects. Those samples are collected before the start of treatment, at the time of first tumor assessment, at the time of first and second disease progression. The subjects are treated according to standard of care.

Clinical data are collected at each sampling time. The primary objective of the study is to identify biological, clinical and tumoral factors associated with tumor response according SOC treatment.

ELIGIBILITY:
Inclusion Criteria:

* Documented new diagnosis of lung cancer by histology or cytology, or lung tumor leading to lung cancer suspicion without diagnosis for which an antineoplastic treatment is indicated
* Indication of a treatment by surgery, chemotherapy, radio-chemotherapy, radiotherapy or targeted therapy as first line of lung cancer treatment
* ability of the subject to follow study procedures
* Age > 18 years
* Subject must have at least one measurable and/or assessable lesion in regard with RECIST 1.1 criteria
* Subject is registered with a social security scheme
* Subject is taken in charge at Pneumology department of Lille UH
* Subject has signed an informed consent form

Exclusion Criteria:

* Patient with a history of treatment by antineoplastic chemotherapy, radio-chemotherapy, radiotherapy or targeted therapy, or presenting a contra indication to antineoplastic treatment administration
* Subject is not willing to sign the informed consent form
* Subject is not registered with a social security scheme
* Subject is not francophone
* Subject is deprived of his/her liberty or under trusteeship

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study includes patients taken in charge at UH Lille, department of pneumology and thoracic oncology (may be also treated at thoracic surgery department, in same hospital). The subjects have a lung cancer diagnosis (all stages are eligible) or a suspicion of lung cancer ; they are included before any treatment initiation.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2019-03-13 (Actual); Primary Completion 2032-03 (Estimated); Study Completion 2032-03 (Estimated)

PRIMARY OUTCOMES:
Objective response rate assessed by CT scan | 8 weeks
  Assessment of tumor response to SOC treatment, using RECIST 1.1 criteria (partial response defined as a decrease of at least 30% in size of target lesions, complete response defined as a disappearance of all lesions)

SECONDARY OUTCOMES:
Disease progression rate assessed by CT scan | 8 weeks
  Assessment of tumor response to SOC treatment, using RECIST 1.1 criteria (disease progression defined as an increasement of at least 20 % in size of target lesions, and/or appearance of new lesions)
Progression-free survival | 8 weeks
Overall survival | 1 year
  number of subjects alive
treatment toxicity | 8 weeks
  length (in days) and grade of the treatment-related toxicities, using Common Terminology Criteria for Adverse Events version 4

OTHER OUTCOMES:
Variation of patient-reported ICEC-R (randomised clinical trials comprehension inventory) | 8 weeks
  This mesure evaluate subject's emotional skills in regard of the clinical trial inclusion process between baseline and first disease assessment (T1), first occurence of progression (T2), second occurence of progression (T3)
Variation of CARE (Consultation and Relational Empathy) questionnaires | 8 weeks
  This mesure evaluate between baseline and first disease assessment (T1), first occurence of progression (T2), second occurence of progression (T3)

CONTACTS AND LOCATIONS:
Overall Officials: Alexis CORTOT, MD,PhD, Principal Investigator — University Hospital, Lille
Locations (1):
- Hôpital Calmette, CHU, Lille, France

IPD SHARING:
Plan to Share IPD: No